CLINICAL TRIAL: NCT03148444
Title: Impact of Antibiotic Treatment Following Implantation of Cardiac Electronic Device on Patient's Outcome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Moshe Swissa, Director, Electrophysiology and Pacing Unit, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: kmc 0038-16
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Infection, Bacterial; Pacemaker Complication
MeSH Terms: conditions — Bacterial Infections | interventions — Cephalexin; Roxithromycin; BID protein, human

STUDY DESIGN:
Intervention Model Description: We propose to organize a randomized open-label study in which patients undergoing de novo implantation or replacement of cardiac implantable devices (single-chamber, dual-chamber and biventricular pacemakers and defibrillators) will be randomly assigned to one of the two groups. Patients in one group will be discharged home with recommendations to take antibiotic treatment for 5 days following the procedure (cefalexin 500 mg qid, or in the presence of beta-lactam sensitivity roxythromycin 150 mg bid) while in the other group no recommendations regarding antibiotic treatment will be given. Both groups will receive antibiotic prophylaxis before the procedure according to the current recommendations. In both groups, the aseptic technique during the procedure will be observed, and proper hygienic measures past the implantation will be taken.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The random assignment will be performed by a researcher from the cardiologic team performing the implantation by means of choosing one of two closed envelopes. The treatment will not be placebo-controlled, and therefore the neither the patients nor the attending physicians will not be blinded to the final results of the assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotics treated (Experimental): Patients undergoing de novo implantation or replacement of cardiac implantable devices (single-chamber, dual-chamber and biventricular pacemakers and defibrillators) in our institution will be discharged home with recommendations to take antibiotic treatment for 5 days following the procedure (cefalexin 500 mg qid, or in the presence of beta-lactam sensitivity roxithromycin 150 mg bid)
  Interventions: Drug: cefalexin 500 mg qid or roxithromycin 150 mg bid
- without Antibiotics Treatment (No Intervention): Patients undergoing de novo implantation or replacement of cardiac implantable devices (single-chamber, dual-chamber and biventricular pacemakers and defibrillators) in our institution will be discharged home with no recommendations regarding antibiotic treatment.

INTERVENTIONS:
Drug: cefalexin 500 mg qid or roxithromycin 150 mg bid — antibiotics treatment for five days following implantation of cardiac device
  Arms: Antibiotics treated

SUMMARY:
Background: Infection of cardiac implantable electronic device including wound and pouch infection, bacteraemia and endocarditis is a common complication of device insertion. The role of antibiotic prophylaxis in prevention of this complication is well established. Most centres in Israel currently prescribe antibiotics about 5 days following the procedure as well, though clear clinical evidence warranting this practise is lacking. Unnecessary antibiotic treatment can lead to adverse events including allergy, undesirable effects of the antibiotics, establishment of resistance to antibiotics among bacteria and further infections with resistant strains.

Objective: The investigators hope to either establish evidence warranting use of post-procedural antibiotic treatment or refuting it.

Methods: The investigators intend to recruit about 400 patients a year into both trial group and control group. The trial group will be treated with post-procedural antibiotics during 5 days, while the control group will receive no post-procedural antibiotics. The endpoints of the study will include infections related to the implantable device and proposed adverse effects of the antibiotics. The t-test will be performed in order to evaluate whether benefit exists concerning one of the groups.

DETAILED DESCRIPTION:
The infection of cardiac implantable electronic device site (including both pocket infection and deeper infections) is a common complication of electronic device insertion. Its incidence is estimated in different series as 0.2-0.7 per 100 device-years. The risk factors that raise the incidence of this complication are in the first place lack of or inappropriate antibiotic prophylaxis and repeated or recurrent manipulations with the device. Several comorbidities such as diabetes, renal insufficiency, heart failure, malignancy, anticoagulation treatment, and, non-surprisingly glucocorticoid treatment are the remaining risk factors for the infection. It is worth mentioning that over half of all cases of infection occur during the first year past implantation.

About 75% of all device infections are caused by staphylococci (both S. aureus and coagulase negative staphylococci). The other causative organisms are streptococci, Corynebacterium species, Propionibacterium, gram-negative bacilli and fungi. Main source of infection appears to be pocket contamination by skin flora. In one study the swab specimens obtained from device pockets during the procedure rendered positive culture for coagulase-negative staphylococci in up to one half of the specimens even despite observant aseptic technique and appropriate antibiotic prophylaxis.Thus, the contamination leading to infection of the implantation site can occur during the procedure. Other possible paths for infection include erosion of the device or its leads through the skin and seeding of the device and its leads by systemic bacteremia. The treatment of this complication usually requires explantation of the infected device, intravenous antibiotic treatment and then implantation of a new device through the non-infected route.

The principal approach to prevent device infection remain aseptic technique during the procedure and appropriate antibiotic prophylaxis. Different clinical trials showed that pre-treatment of elective patients before the device implantation with anti-staphylococcal penicillins or with first generation cephalosporins results in decrease in rate of infection with odds ratio about 0.2-0.25.Therefore, current recommendation is to pre-treat patients before implantation of the device with 2-3 gram cefazolin or 1.5 gram cefuroxime, or 15 mg/kg vancomycin or clindamycin 900 mg IV within 4 hours before the procedure. Currently there is no evidence regarding adjuvant antibiotic treatment after the implantation. In the face of lack of evidence, several medical centres in Israel either non-uniformly administer different antibiotic regimens following the implantation or refrain from routinely prescribing any antibiotics to the patients following the implantation.

Objective:

The investigators suppose that non-necessary antibiotic treatment entails several adverse outcomes including direct adverse effects of the antibiotics (e.g. allergy, gastrointestinal effects, QT-prolongation), and induction of resistance to antibiotics among the patient's microflora entailing further infections with resistant bacteria (e.g. urinary tract infections, diarrhea). Therefore, an evidence either warranting use of antibiotics following the implantation of implantable electronic device or refuting it should be established.

Medications:

1. cefalexin 500 mg qid,
2. roxithromycin 150 mg bid Both medications are authorized in Israel for a variety of infections or infection prevention including prevention of implantable cardiac electronic device infection. Both medications are routinely prescribed in medical centres in Israel following implantation of cardiac electronic devices.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing de novo implantation or replacement of cardiac implantable devices (single-chamber, dual-chamber and biventricular pacemakers and defibrillators) in our institution.

Exclusion Criteria:

* procedure during which, according to the opinion of the operator, the risk of the contamination would be unusually high (for ex. due to prolonged duration) so that obligatory post-operative use of antibiotics should be warranted,
* patients with any immunosuppressive condition (including cytotoxic chemotherapy, chronic use of glucocorticoids, however excluding diabetes mellitus, renal failure and heart failure);
* malignancy,
* pregnancy and breastfeeding;
* hepatic cirrhosis;
* end stage renal disease (GFR<10 mL/min);
* known allergy to both antibiotic medications used in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
wound infection | 1 year
  operative wound infection or infection of the device pouch
bacteremia and vegetations | 1 year
  bacteremia due to device infection, lead vegetation, right infective endocarditis
re-operation | 1 year
  re-operation due to infective complications

SECONDARY OUTCOMES:
infection unrelated to implantation | 1 year
  any infection (e.g. bacteremia, urinary tract infection, diarrhea) unrelated to the implantable device, whether demanding hospitalization or not
hospitalization | 1 year
  any hospitalization due to non-infective problems related to the implantable device
adverse event of antibiotics | 1 year
  any event related to adverse effect of antibiotics warranting discontinuation of the drug e.g. allergy
death from any cause | 1 year
  death from any cause unrelated to the problems enumerated among primary outcomes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Uslan DZ, Sohail MR, St Sauver JL, Friedman PA, Hayes DL, Stoner SM, Wilson WR, Steckelberg JM, Baddour LM. Permanent pacemaker and implantable cardioverter defibrillator infection: a population-based study. Arch Intern Med. 2007 Apr 9;167(7):669-75. doi: 10.1001/archinte.167.7.669. PMID 17420425
- [Background] Klug D, Balde M, Pavin D, Hidden-Lucet F, Clementy J, Sadoul N, Rey JL, Lande G, Lazarus A, Victor J, Barnay C, Grandbastien B, Kacet S; PEOPLE Study Group. Risk factors related to infections of implanted pacemakers and cardioverter-defibrillators: results of a large prospective study. Circulation. 2007 Sep 18;116(12):1349-55. doi: 10.1161/CIRCULATIONAHA.106.678664. Epub 2007 Aug 27. PMID 17724263
- [Background] Smith PN, Vidaillet HJ, Hayes JJ, Wethington PJ, Stahl L, Hull M, Broste SK. Infections with nonthoracotomy implantable cardioverter defibrillators: can these be prevented? Endotak Lead Clinical Investigators. Pacing Clin Electrophysiol. 1998 Jan;21(1 Pt 1):42-55. doi: 10.1111/j.1540-8159.1998.tb01060.x. PMID 9474647
- [Background] Da Costa A, Lelievre H, Kirkorian G, Celard M, Chevalier P, Vandenesch F, Etienne J, Touboul P. Role of the preaxillary flora in pacemaker infections: a prospective study. Circulation. 1998 May 12;97(18):1791-5. doi: 10.1161/01.cir.97.18.1791. PMID 9603533
- [Background] Da Costa A, Kirkorian G, Cucherat M, Delahaye F, Chevalier P, Cerisier A, Isaaz K, Touboul P. Antibiotic prophylaxis for permanent pacemaker implantation: a meta-analysis. Circulation. 1998 May 12;97(18):1796-801. doi: 10.1161/01.cir.97.18.1796. PMID 9603534
- [Background] de Oliveira JC, Martinelli M, Nishioka SA, Varejao T, Uipe D, Pedrosa AA, Costa R, D'Avila A, Danik SB. Efficacy of antibiotic prophylaxis before the implantation of pacemakers and cardioverter-defibrillators: results of a large, prospective, randomized, double-blinded, placebo-controlled trial. Circ Arrhythm Electrophysiol. 2009 Feb;2(1):29-34. doi: 10.1161/CIRCEP.108.795906. Epub 2009 Feb 10. PMID 19808441
- [Background] Sohail MR, Uslan DZ, Khan AH, Friedman PA, Hayes DL, Wilson WR, Steckelberg JM, Stoner S, Baddour LM. Management and outcome of permanent pacemaker and implantable cardioverter-defibrillator infections. J Am Coll Cardiol. 2007 May 8;49(18):1851-9. doi: 10.1016/j.jacc.2007.01.072. Epub 2007 Apr 23. PMID 17481444
- [Background] Lekkerkerker JC, van Nieuwkoop C, Trines SA, van der Bom JG, Bernards A, van de Velde ET, Bootsma M, Zeppenfeld K, Jukema JW, Borleffs JW, Schalij MJ, van Erven L. Risk factors and time delay associated with cardiac device infections: Leiden device registry. Heart. 2009 May;95(9):715-20. doi: 10.1136/hrt.2008.151985. Epub 2008 Nov 26. PMID 19036758